CLINICAL TRIAL: NCT07079644
Title: Real World Outcomes of Nivolumab + Relatlimab in Patients With Advanced Melanoma in the Flatiron Database
Brief Title: Outcomes of Nivolumab in Combination With Relatlimab in Patients With Advanced Melanoma in the Flatiron Database
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA224-1098
Record Dates: First submitted 2025-06-10; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Advanced Melanoma
Keywords: Advanced melanoma
MeSH Terms: interventions — Nivolumab; relatlimab; Ipilimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1L Nivolumab + Relatlimab cohort
  Interventions: Biological: Nivolumab + Relatlimab
- 1L Nivolumab + Ipilimumab cohort
  Interventions: Biological: Nivolumab + Ipilimumab
- 1L Immunotherapy monotherapy cohort
  Interventions: Biological: Immunotherapy monotherapy
- 1L BRAF/MEKs inhibitors cohort
  Interventions: Drug: BRAF/MEK inhibitors

INTERVENTIONS:
Biological: Nivolumab + Relatlimab — As per product label
  Groups: 1L Nivolumab + Relatlimab cohort
Biological: Nivolumab + Ipilimumab — As per product label
  Groups: 1L Nivolumab + Ipilimumab cohort
Biological: Immunotherapy monotherapy — As per product label
  Groups: 1L Immunotherapy monotherapy cohort
Drug: BRAF/MEK inhibitors — As per product label
  Groups: 1L BRAF/MEKs inhibitors cohort

SUMMARY:
The purpose of this study is to investigate the real-world clinical outcomes of individuals that have been diagnosed with advanced melanoma who were treated with Nivolumab in combination with Relatlimab, Nivolumab in combination with Ipilimumab, immuno-oncology monotherapy or BRAF/MEK inhibitors therapy

ELIGIBILITY:
Inclusion Criteria:

* Participants in the advanced melanoma cohort

  * Participants included in the cohort by Flatiron criteria of: cutaneous melanoma with pathologic stages III or IV, either at initial diagnosis or via local or distant recurrence, and at least two clinic encounters evident in the database
* Participants receiving Nivolumab + Relatlimab between March 18, 2022 and September 30, 2024 or other therapies (Nivolumab + Ipilimumab, immunotherapy monotherapy, BRAF/MEK inhibitors) between March 18, 2022 and November 30, 2024 (or date of the most recent data cut off)
* Participants ≥18 years old on index date
* Participants with ≥1 month of medical data after the index date (inclusive), unless patient died within this period

Exclusion Criteria:

* Participants with diagnosis of other primary cancers prior to the index date
* Participants receiving medication in a clinical trial at any time prior to, on or after index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adults identified from the Flatiron database that have been diagnosed with advanced melanoma and who have initiated treatment with either Nivolumab in combination with Relatlimab, Nivolumab in combination with Ipilimumab, immuno-oncology monotherapy or BRAF/MEK inhibitors therapy in the real-world clinical settings
Sampling Method: Non-Probability Sample
Enrollment: 678 (Actual)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Demographics | Baseline
Clinical characteristics: Location of metastatic sites | Baseline
Clinical characteristics: Lactate dehydrogenate (LDH) test results | Baseline
Clinical characteristics: BRAF status | Baseline
Clinical characteristics: Eastern Cooperative Oncology Group Performance Status (ECOG PS) | Baseline
Overall survival (OS) | Up to 3-years
Real-world progression-free survival (rwPFS) | Up to 3-years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol Myers Squibb, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts